CLINICAL TRIAL: NCT03197909
Title: Involvement of Plasmatic Factors in the Peripheral Muscle Dysfunction of COPD Patients - In Vitro Study
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0210
Record Dates: First submitted 2017-06-21; First posted 2017-06-23 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2018-09

CONDITIONS: Chronic Obstructive Pulmonary
Keywords: COPD (Chronic Obstructive Pulmonary Patients); Atrophy; cell cultur; systemic inflammation; Catabolism
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Atrophy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy subjects: Determination of pro-inflammatory plasma factors at Healthy subjects aged from 35 to 85 years old
  Interventions: Other: Determination of pro-inflammatory plasma factors
- COPD patients: Determination of pro-inflammatory plasma factors at COPD patients aged from 35 to 85 years old
  Interventions: Other: Determination of pro-inflammatory plasma factors

INTERVENTIONS:
Other: Determination of pro-inflammatory plasma factors — Determination of pro-inflammatory plasma factors at COPD patients aged from 35 to 85 years old and Healthy subjects aged from 35 to 85 years old

SUMMARY:
Chronic Obstructive Pulmonary Patients is a defined by persistent airflow limitation that is usually progressive and associated with an enhanced chronic inflammatory response in the airways and the lung to noxious particles or gases. It is associated with an atrophy of the skeletal muscle that impairs the patient's prognosis. The biological mechanisms of this muscle atrophy have not been elucidated, and the "spill-over theory" has recently emerged. Indeed, in COPD patients, the pulmonary inflammation is associated with a systemic low-grade inflammation, and the increased pro-inflamatory molelcules in the blood - which constitute the cellular micro-environement of the muscle fibre - could activate the mechanisms of the cell atrophy.

ELIGIBILITY:
Inclusion Criteria:

35 to 85 years old

* COPD patients: association of symtoms (breathlessness, cough, sputum) and chronic exposure to inhalated risk factors (like tobacco smoke) and a FEV1/VC ratio <70% assessed by a spirometry
* Healthy subjects: A sedentariness assessed by a Voorrips score <9.4 and/or a report of <150 min/week of moderate-to-vigorous physical activity

Exclusion Criteria:

* A recent COPD exacerbation (< 4weeks)
* The decompensation of a comorbidity
* An antioxidant supplementation or medication
* A long-term systemic corticosteroid medication

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Chronic Obstructive Pulmonary Patients
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2017-07-06 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-01-31 (Actual)

PRIMARY OUTCOMES:
Myotube diameter of in vitro cultured myotubes | 6 days
  Myotube diameter of in vitro cultured myotubes from healthy subjects, exposed to the serum of healthy controls and COPD patients

SECONDARY OUTCOMES:
Expression and translation of markers of | 6 days
  Expression and translation of markers of anabolic and catabolic pathways

OTHER OUTCOMES:
Level of pro-Inflamatory markers | 6 days
  Level of pro-Inflamatory markers in the serum

CONTACTS AND LOCATIONS:
Overall Officials: Maurice HAYOT, MD, PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC